CLINICAL TRIAL: NCT02052830
Title: Impact Evaluation of the Wise Guys Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRP699101
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2015-09

CONDITIONS: Sexual Behavior; Sexually Transmitted Infections
MeSH Terms: conditions — Sexual Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wise Guys (Experimental): A sexual health and male responsibility program for adolescent males
  Interventions: Behavioral: Wise Guys
- Control (No Intervention): Business as usual sexual education in schools

INTERVENTIONS:
Behavioral: Wise Guys — Multi-session curriculum delivered in different formats that range in length from 5 to 12 weeks and topics covered include communication and masculinity, dating violence, abstinence and contraception, and sexually transmitted infections.
  Arms: Wise Guys

SUMMARY:
The purpose of this study is to evaluate the impact of the Wise Guys program on the delaying sexual initiation on adolescent males in Eastern Iowa.

DETAILED DESCRIPTION:
This study uses a randomized controlled design to compare the impacts of the Wise Guys Program to the "business-as-usual" school curriculum. The Wise Guys multi-session curriculum is delivered in different formats that range in length from 5 to 12 weeks and topics covered include communication and masculinity, dating violence, abstinence and contraception, and sexually transmitted infections. Study participants are 7th grade boys attending a participating school in either the Davenport Iowa or North Scott Community school districts. This study is being conducted as part of the national Personal Responsibility Education Program evaluation funded by Administration for Children and Families within the U.S. Department of Health and Human Services.

ELIGIBILITY:
Inclusion Criteria:

* 7th grade student in participating schools
* Male

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Sexual initiation | 24 months post-intervention

SECONDARY OUTCOMES:
Sexual initiation | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, PhD, Study Director — Mathematica Policy Research